CLINICAL TRIAL: NCT06785155
Title: AI Chatbot-Based Learning on Dry Eye and Eye Strain Knowledge Among Nursing Students
Brief Title: AI Chatbot-Based Learning on Dry Eye and Eye Strain Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, İbrahim Edhem Yılmaz, Assistant Professor, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GaziantepIslamSTU-01
Record Dates: First submitted 2025-01-09; First posted 2025-01-21 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Health Behaviors; Artificial Intelligence (AI); Chatbot; Dry Eye; Eye Strain
MeSH Terms: conditions — Health Behavior; Dry Eye Syndromes; Asthenopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- website group (Active Comparator): Participants explored these topics using the website.
  Interventions: Other: website assisted
- Chatbot group (Experimental): Participants explored the topics using the AI chatbot platform
  Interventions: Other: Chatbot group

INTERVENTIONS:
Other: Chatbot group — Participants explored the topics using the AI chatbot platform.
  Arms: Chatbot group
Other: website assisted — Participants explored the topics using the website platform
  Arms: website group

SUMMARY:
The aim of this project is to evaluate the effectiveness of using chatbots for patient education about dry eye disease. The study will examine how the chatbot affects patients' levels of information, managing symptoms, and overall satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* to be actively enrolled in the nursing program
* to demonstrate baseline digital literacy.

Exclusion Criteria:

* diagnosed visual impairments,
* those with prior specialized ophthalmological training,
* individuals with limited digital technology proficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Dry Eye and eye strain knowledge questionnaire | From enrollment to the end of training at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Deparment of Nursing, Kilis 7 Aralık University, Kilis, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No